CLINICAL TRIAL: NCT06431815
Title: Prospective, Multi-site Safety and Effectiveness Post-Approval Study of FARAPULSE Pulsed Field Ablation in Paroxysmal Atrial Fibrillation
Brief Title: ADVENT Post Approval Study
Acronym: ADVENTPAS
Status: Active, not recruiting | Type: Observational
Sponsor: Boston Scientific Corporation (Industry)
Responsible Party: Sponsor
Other Study IDs: PF304
Record Dates: First submitted 2024-05-22; First posted 2024-05-29 (Actual); Last update posted 2026-01-28 (Actual); Status verified 2026-01

CONDITIONS: Paroxysmal Atrial Fibrillation
Keywords: Pulsed Field Ablation; PFA; Pulmonary Vein Isolation; PVI; Ablation; Atrial Fibrillation; AF
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

INTERVENTIONS:
Device: FARAPULSE™ Pulsed Field Ablation System — De-novo pulmonary vein isolation (PVI) will be performed with the FARAPULSE Pulsed Field Ablation (PFA) System.
  Other Names: FARAWAVE™ Pulsed Field Ablation Catheter

SUMMARY:
The ADVENT Post Approval Study (PAS) is a prospective, global, multicenter, observational study.

DETAILED DESCRIPTION:
The objective of ADVENT PAS is to evaluate the long-term safety and effectiveness profile of the FARAPULSE Pulsed Field Ablation System when used to perform pulmonary vein isolation (PVI) in the de-novo ablation treatment of patients with paroxysmal atrial fibrillation (PAF).

ELIGIBILITY:
Inclusion Criteria:

* Subjects with drug-refractory, recurrent, symptomatic paroxysmal atrial fibrillation (PAF) who are indicated for a treatment with the FARAPULSE Pulsed Field Ablation (PFA) System*; (Subjects refractory, or intolerant or contraindicated to at least one class I or III antiarrhythmic medication or contraindicated to any class I or III medications.)
* Subjects who are willing and capable of providing informed consent;
* Subjects who are willing and capable of participating in all testing and follow-up associated with this clinical study at an approved clinical investigational site;
* Subjects who are of legal age to give informed consent specific to the national law.
* For the LUX-Dx Sub-Study: Subjects with an existing LUX-Dx Insertable Cardiac Monitor (ICM), inserted ≥ 180 days prior to enrollment, or having a LUX-Dx ICM inserted per the investigator's standard of care, up to 7 days after the ablation procedure. Subjects with or having a LUX-Dx ICM inserted per standard of care, up to 7 days after the ablation procedure.

Exclusion Criteria:

* Subjects with any known contraindication to an AF ablation or anticoagulation, including those listed in the Instructions For Use (IFU);
* Subjects with any prior left atrium (LA) ablation;
* Subjects who may need an ablation in the left atrium besides PVI, such as for left-sided atrioventricular reentrant tachycardia (AVRT), left-sided atrial tachycardia (AT) or atypical left-sided atrial flutter (AFL);
* Women of childbearing potential who are or plan to become pregnant during the time of the study (assessment per investigator's discretion);
* Life expectancy of < 1 year, per investigator's medical judgement.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects with drug-refractory, recurrent, symptomatic paroxysmal atrial fibrillation (PAF) who are indicated for a de-novo pulmonary vein isolation ablation with the FARAPULSE Pulsed Field Ablation (PFA) System.
Sampling Method: Non-Probability Sample
Enrollment: 228 (Actual)
Dates: Start 2024-09-25 (Actual); Primary Completion 2028-10 (Estimated); Study Completion 2029-10 (Estimated)

PRIMARY OUTCOMES:
Composite incidence of patients with procedure-related and device-related serious adverse events at 7-Days and 12-months post-Index Procedure. | 12 Months
  * Early Onset: Acute primary safety endpoint events, events occurring up to 7 days post-Index Procedure or hospital discharge, whichever is later including serious procedure-related and device-related adverse events.
    * Death
    * Myocardial infarction (MI)
    * Persistent phrenic nerve palsy
    * Stroke/Cerebrovascular accident (CVA)
    * Transient ischemic attack (TIA)
    * Peripheral or organ thromboembolism
    * Cardiac tamponade / perforation
    * Pericarditis
    * Pulmonary edema
    * Serious vascular access complications
    * Heart block
    * Gastric motility / pyloric spasm disorders
    * Severe hemolysis with subsequent renal injury or significant anemia
  * Late Onset: Either of the following with an onset date any time through 12-month post-Index Procedure:
  * Atrial esophageal fistula
  * Pulmonary vein stenosis (≥ 70% reduction of diameter)
Treatment success, defined as the incidence of subjects with successful isolation of clinically relevant pulmonary veins AND patients without recurrence or interventions for AF, AFL, AT after the blanking period through 12 months. | 12 Months
  - Acute Procedural Success: Acute procedural success is defined as isolation of all clinically relevant pulmonary veins or anatomical equivalents using the FARAPULSE Pulsed Field Ablation System only
  AND
  - Chronic Success, defined as freedom from the following:
  After the Blanking Period up to the 12-Month Follow-up visit:
  * Occurrence of any Detectable AF, AFL, AT
  * ≥ 30 seconds in duration from any approved clinical recording devices considered standard of care at the study center (excluding implantable loop recorders) or
  * ≥ 10-second of continuous AF, AFL or AT documented on any 12-lead ECG
  * Following interventions:
  * Any cardioversion for AF, AFL or AT
  * Prescribed a higher dose of any failed Class I or III Antiarrhythmic Drug (AAD) documented at baseline or any new Class I or III AAD
  * Re-ablation for AF, AFL or AT (other than for cavotricuspid isthmus (CTI)-dependent flutter only)

CONTACTS AND LOCATIONS:
Overall Officials: Stavros E Mountantonakis, MD, MBA, Principal Investigator — Northwell Health, Lenox Hill Hospital
Locations (30):
- United States (25):
  - Mobile Infirmary Medical Center, Mobile, Alabama
  - Scottsdale Healthcare - Shea, Scottsdale, Arizona
  - Alta Bates Summit Medical Center, Oakland, California
  - Washington Hospital Center, Washington D.C., District of Columbia
  - Florida Heart Rhythm Specialists, PLLC, Fort Lauderdale, Florida
  - Baptist Medical Center, Jacksonville, Florida
  - Mount Sinai Medical Center, Miami Beach, Florida
  - Tallahassee Memorial Hospital, Tallahassee, Florida
  - AdventHealth Tampa, Tampa, Florida
  - Memorial Health University Medical Center, Savannah, Georgia
  - Ochsner Clinic Foundation, New Orleans, Louisiana
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - University of Mississippi Medical Center, Jackson, Mississippi
  - New York Hospital Queens, Flushing, New York
  - Columbia University Medical Center, New York, New York
  - Northwell Health, New York, New York
  - Montefiore Medical Center, The Bronx, New York
  - East Carolina University Medical Center, Greenville, North Carolina
  - Pinnacle Health at Harrisburg Hospital, Harrisburg, Pennsylvania
  - Medical University of South Carolina, Charleston, South Carolina
  - Prisma Health Richland Hospital, Columbia, South Carolina
  - University of Texas Medical Branch, Galveston, Texas
  - University of Texas Houston Health Science Center, Houston, Texas
  - Orion Medical, Houston, Texas
  - Sentara Norfolk General Hospital, Norfolk, Virginia
- Brazil (2):
  - Sos Cardio Servicoshospitalares Ltda, Florianópolis, Santa Catarina
  - Instituto do Coração do HCFMUSP, São Paulo, São Paulo
- Canada (2):
  - Institut de Cardiologie de Montreal-Hospital, Montreal, Quebec
  - Institut universitaire de Cardiologie et de Pneumologie de Quebec, Québec, Quebec
- Hospital Regional de Concepcion, Concepción, Región del Biobío, Chile

IPD SHARING:
Plan to Share IPD: Undecided
No requests for study data have been made at this time, however Boston's Scientific's policy on data sharing can be found at http://www.bostonscientific.com/en-US/data-sharing-requests.html